CLINICAL TRIAL: NCT04019366
Title: Effects of Balance Training Using Biodex Stability System in Patients With Symptomatic Knee Osteoarthritis.
Brief Title: Balance Training Using Biodex Stability System in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Samina Javed
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: Balance Training; Biodex stability system; Osteoarthrosis; Degenerative; Stability exercises
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment of patients into two groups
Who Masked: Participant
Masking Description: Patients were masked from the treatment procedure by Sealed envelope methods. Patients were randomly distributed into two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): The experimental group was treated with Balance Training on Biodex Stability System along with traditional exercises.
  Interventions: Other: Balance Training
- Group II (Active Comparator): The Control group was treated with Traditional exercises only for Symptomatic knee osteoarthritis.
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Balance Training — Experimental group received balance training on Biodex stability System along with traditional exercise program. During balance training on Biodex, patients were instructed to stand on the platform with bare feet with open eyes and both legs supported. Patients were looking forward to screen having hands hang by the sides. The patients were instructed not to change their feet position and balance the body. The handles were accessible for safety point. But touching the handles cancelled the trail. Total time of training was 10 minutes each set is of 3 minutes with 20 sec rest intervals.
  Arms: Group I
Other: Conventional Training — Control group has received traditional exercises i.e Quadriceps strength exercises, Hamstrings flexibility exercises and Balance exercises.
  Arms: Group II

SUMMARY:
This was a randomized control Trial, conducted with two group of patients, one has received Balance and stability training on Biodex stability system along with conservative protocol of traditional exercises. the other group has received only conservative protocol of traditional exercises

DETAILED DESCRIPTION:
Patients with Symptomatic Knee Osteoarthritis have balance and stability deficits. In routine such patients are not evaluated and treated on balance and stability parameters. So this study was conducted with objectives to determine the effects of Balance training using Biodex stability system in patients with symptomatic knee osteoarthritis.

Experimental group has received Balance and stability training on Biodex stability system along with conservative protocol of traditional exercises.

Control group has received only conservative protocol of traditional exercises.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral knee pain
* Age 35-65, Both genders
* Grade 2 or 3 on Kellgren classification for Knee Arthritis

Exclusion Criteria:

* Past history of total knee artthroplasty
* Intra articular steroid injection
* Rheumatoid Arthritis
* Use of Assistive devices e.g. canes, walkers and braces
* Knee injury

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Time up and Go test (TUG) | Baseline
  Patients were asked to perform test at usual walking speed. Initial testing standardized verbal instructions given to the participant regarding procedure. For performing TUG participants were instructed to walk three meter and then, walk back to sit down. Note time on stopwatch. The average of tests trail was measured as the mean of TUG.
Time up and Go test (TUG) | Post 4th Week
  Patients were asked to perform test at usual walking speed. Initial testing standardized verbal instructions given to the participant regarding procedure. For performing TUG participants were instructed to walk three meter and then, walk back to sit down. Note time on stopwatch. The average of tests trail was measured as the mean of TUG.
overall stability index (OSI) | Baseline
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .94
overall stability index (OSI) | Post 4th Week
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .94
Anterior-posterior stability index (APSI) | Baseline
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .95
Anterior-posterior stability index (APSI) | Post 4th Week
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .95
Medial-lateral stability index (MLSI) | Baseline
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .93
Medial-lateral stability index (MLSI) | Post 4th Week
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .93

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric Pain Rating Scale (NPRS) | post 4th week
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline
  It is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items):Stiffness (2 items): Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Post 4th week
  It is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items):Stiffness (2 items): Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Armed forces Institute of Rehabilitation Medicine (AFIRM), Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldwin SL, Das JP. Atmospheric Ar and Ne returned from mantle depths to the Earth's surface by forearc recycling. Proc Natl Acad Sci U S A. 2015 Nov 17;112(46):14174-9. doi: 10.1073/pnas.1424122112. Epub 2015 Nov 5. PMID 26542683
- [Background] Huang MH, Lin YS, Yang RC, Lee CL. A comparison of various therapeutic exercises on the functional status of patients with knee osteoarthritis. Semin Arthritis Rheum. 2003 Jun;32(6):398-406. doi: 10.1053/sarh.2003.50021. PMID 12833248
- [Background] Chuang SH, Huang MH, Chen TW, Weng MC, Liu CW, Chen CH. Effect of knee sleeve on static and dynamic balance in patients with knee osteoarthritis. Kaohsiung J Med Sci. 2007 Aug;23(8):405-11. doi: 10.1016/S0257-5655(07)70004-4. PMID 17666307
- [Background] Eftekhar-Sadat B, Azizi R, Aliasgharzadeh A, Toopchizadeh V, Ghojazadeh M. Effect of balance training with Biodex Stability System on balance in diabetic neuropathy. Ther Adv Endocrinol Metab. 2015 Oct;6(5):233-40. doi: 10.1177/2042018815595566. PMID 26445646